CLINICAL TRIAL: NCT04088396
Title: Open-Label, Randomized Study With a Tocilizumab Reference Arm to Evaluate Safety, Efficacy and Pharmacokinetics of Baricitinib in Children From 1 to Less Than 18 Years of Age With Systemic Juvenile Idiopathic Arthritis.
Brief Title: A Study of Baricitinib (LY3009104) in Participants From 1 Year to Less Than 18 Years Old With Systemic Juvenile Idiopathic Arthritis (sJIA)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16275; I4V-MC-JAHU (Other: Eli Lilly and Company); 2017-004495-60 (EudraCT Number); 2023-507883-38-00 (EU CTIS Number)
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Systemic Juvenile Idiopathic Arthritis
Keywords: Systemic; Fever; Flare; sJIA; JIA
MeSH Terms: conditions — Arthritis, Juvenile; Fever | interventions — baricitinib; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 Baricitinib (Experimental): Baricitinib given orally.
  Interventions: Drug: Baricitinib
- Cohort 1 Tocilizumab (Active Comparator): Tocilizumab given Subcutaneously (SC).
  Interventions: Drug: Tocilizumab
- Cohort 2 Baricitinib (Experimental): Baricitinib given orally.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
  Arms: Cohort 1 Baricitinib; Cohort 2 Baricitinib
Drug: Tocilizumab — Administered SC
  Arms: Cohort 1 Tocilizumab

SUMMARY:
The reason for this study is to see if the study drug baricitinib is safe and effective in participants from 1 year to less than 18 years old with systemic juvenile idiopathic arthritis (sJIA). Participants are assigned to 1 of 2 cohorts. In cohort 1, participants will receive baricitinib or tocilizumab reference. In cohort 2, participants will receive baricitinib.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of systemic Juvenile Idiopathic Arthritis (sJIA) as defined by International League of Associations for Rheumatology (ILAR) criteria with onset before the age of 16 years
* Participants must have at least 2 active joints at screening and baseline
* Cohort 1 (IL-6 inhibitor therapy naive): Participants who are at least 1 year and less than 18 years of age, except in countries that restrict use of tocilizumab in participants less than 2 years of age
* Cohort 2 (open-label baricitinib): Participants who are at least 1 year and less than 18 years of age

Exclusion Criteria:

* Participants must not have polyarticular JIA (positive or negative for rheumatoid factor), extended oligoarticular JIA, enthesitis-related JIA, or juvenile psoriatic arthritis
* Participants must not have persistent oligoarticular arthritis as defined by the ILAR criteria
* Participants must not have a history or presence of any autoimmune inflammatory condition other than JIA
* Participants must not have active anterior uveitis or are receiving concurrent treatment for anterior uveitis
* Participants must not have active fibromyalgia or other chronic pain conditions that, in the investigator's opinion, would make it difficult to appropriately assess disease activity for the purposes of this study
* Participants must not have biologic features of Macrophage Activation Syndrome (MAS) over the past 12 weeks
* Participants must not have a current or recent (<4 weeks prior to baseline) clinically serious infection
* Participants must not have a positive test for hepatitis B virus
* Participants must not have evidence of active tuberculosis (TB) or untreated latent TB

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Adapted Pediatric American College of Rheumatology 30 Responder Index (PediACR30) Response Criteria at Week 12 | Week 12
  Percentage of Participants Achieving Adapted PediACR30 Response Criteria

SECONDARY OUTCOMES:
Percentage of Participants Achieving Adapted PediACR30 Response Criteria at Week 24 | Week 24
  Percentage of Participants Achieving Adapted PediACR30 Response Criteria
Percentage of Participants with Inactive Disease | Week 12
  Percentage of Participants with Inactive Disease
Percentage of Participants with Minimal Disease Activity | Week 12
  Percentage of Participants with Minimal Disease Activity
Change from Baseline in Juvenile Arthritis Disease Activity Score (JADAS)-27 | Baseline, Week 24
  Change from Baseline in JADAS-27
Change from Baseline in Arthritis-Related Pain Severity as Measured by the Childhood Health Assessment Questionnaire (CHAQ) Pain Visual Analog Scale (VAS) Item | Baseline, Week 24
  Change from Baseline in Arthritis-Related Pain Severity as Measured by the CHAQ Pain VAS Item
Pharmacokinetics (PK): Maximum Plasma Baricitinib Concentration at Steady-State (Cmax, ss) | Baseline through Week 24
  PK: Cmax, ss of Baricitinib
PK: Area Under the Baricitinib Concentration-Time Curve at Steady-State (AUC, ss) | Baseline through Week 24
  PK: AUC, ss of Baricitinib

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (55):
- Argentina (2):
  - Instituto CAICI SRL, Rosario
  - Centro Medico Privado de Reumatologia, SAN M. de Tucuman
- UZ Gent, Ghent, Belgium
- Brazil (5):
  - Faculdade de Medicina da UNESP, Botucatu
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - IPITEC, São Paulo
  - Universidade Federal de Sao Paulo, São Paulo
  - Instituto da Crianca do Hospital das Clinicas da FMUSP, São Paulo
- Czechia (2):
  - Detska nemocnice FN Brno, Brno
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (5):
  - Hospices Civils de Lyon - Hôpital Femme Mère Enfant, Bron
  - Hôpitaux Universitaires Paris Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier Universitaire de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - Hôpital Universitaire Necker Enfants Malades, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
- Sir Ganga Ram Hospital, New Delhi, India
- Israel (3):
  - Meir Medical Center, Kfar Saba
  - Schneider Children's Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Italy (8):
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Azienda Sanitaria Locale n. 2 - Lanciano Vasto Chieti, Chieti
  - IRCCS Istituto Giannina Gaslini, Genova
  - Centro Specialistico Ortopedico Traumatologico Gaetano Pini - CTO, Milan
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - University of Naples Federico II, Napoli
  - Azienda di Rilievo Nazionale e Alta Specializzazione Civico Di Cristina Benfratelli, Palermo
  - Ospedale Infantile Burlo Garofolo, Trieste
- Japan (7):
  - Institute of Science Tokyo Hospital, Bunkyō
  - Chiba Children's Hospital, Chiba
  - Kagoshima University Hospital, Kagoshima
  - Miyagi Children's Hospital, Sendai
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki
  - Kanagawa Children's Medical Center, Yokohama
  - Yokohama City University Hospital, Yokohama
- Mexico (5):
  - Investigacion y Biomedicina de Chihuahua, Chihuahua City
  - Instituto de Investigaciones Clínicas para la Salud, Durango
  - Crea de Guadalajara, Guadalajara
  - Clinstile, S.A. de C.V., México
  - Hospital Universitario Dr. José Eleuterio González, Universidad Autónoma de Nuevo León, Monterrey
- Poland (3):
  - Wojewódzki Specjalistyczny Szpital Dziecięcy im. św. Ludwika w Krakowie, Krakow
  - Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi, Lodz
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji, Warsaw
- Spain (6):
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Turkey (Türkiye) (2):
  - Istanbul University-Cerrahpasa, Cerrahpasa Faculty of Medicine, Istanbul
  - 9 Eylul University Hospital, Izmir
- United Kingdom (5):
  - Bristol Royal Hospital for Children, Bristol
  - Alder Hey Children's Hospital, Liverpool
  - Great Ormond Street Hospital For Children NHS Foundation Trust, London
  - Oxford University Hospitals - Nuffield Orthopaedic Centre, Oxford
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://www.vivli.org/

REFERENCES:
- See also: A Study of Baricitinib (LY3009104) in Participants From 1 Year to Less Than 18 Years Old With sJIA — https://trials.lillytrialguide.com/en-US/trial/4qr6645c2hmeJZWASkU2jH